CLINICAL TRIAL: NCT05814159
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Efficacy and Safety Study of Subcutaneous Anakinra in Japanese Patients With Still's Disease (SJIA and AOSD)
Brief Title: A Study of Anakinra in Japanese Patients With Still's Disease (SJIA and AOSD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sobi.ANAKIN-303
Record Dates: First submitted 2022-11-22; First posted 2023-04-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Still's Disease, Juvenile Onset; Still's Disease, Adult-Onset
MeSH Terms: conditions — Arthritis, Juvenile; Still's Disease, Adult-Onset | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anakinra (Experimental): 100 mg/day or 2 mg/kg/day of subcutaneous anakinra for those with a body weight ≥50 kg or <50 kg, respectively.
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Corresponding volume to 100 mg/day or 2 mg/kg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — sub cutaneous daily injection
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — sub cutaneous daily injection
  Arms: Placebo

SUMMARY:
A study to demonstrate efficacy and safety of anakinra in pediatric and adult Japanese patients with Still's disease (Systemic juvenile idiopathic arthritis [SJIA] and Adult-onset Still's disease [AOSD]).

DETAILED DESCRIPTION:
The study consists of two phases:

• Core phase comprising 2 weeks double blind placebo-controlled treatment, 52 weeks open label treatment and 4 weeks safety follow up (only for patients not entering the extension phase).

At the Week 54 visit, patients who consent and are eligible to continue anakinra treatment, will enter the extension phase and continue open label anakinra treatment.

• Extension phase comprising up to 26 weeks open label treatment and 4 weeks safety follow up.

The primary endpoint will be evaluated at Week 2 visit.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female patients, 8 months of age or older with a body weight ≥ 10 kg
2. Diagnosis of Still's disease
3. If < 16 years of age at disease onset, the diagnosis is madeaccording to adapted ILAR criteria i.e., CARRA criteria for SJIA. If ≥ 16 years of age at disease onset, the diagnosis is made according to Yamaguchi criteria for AOSD.
4. Active disease confirmed by the following three signs and symptoms. a. Active arthritis in ≥ 1 joint. b. CRP > 30 mg/L. c. At least one fever episode (≥ 38.0 degree Celsius) attributable to the disease within one week before enrollment.
5. The result of tuberculosis test within 8 weeks prior to enrollment is negative.

Key Exclusion Criteria:

1. Previous or current treatment with anakinra, or any other Interleukin-1 (IL-1) inhibitor except for canakinumab. Previous treatment with canakinumab is allowed if canakinumab was discontinued for reasons other than lack of efficacy and after a washout period of minimum 130 days. Patients who have discontinued canakinumab because of insufficient effect or refractory disease are not allowed to be enrolled in the study.
2. Use of the following therapies prior to enrollment.

   1. Narcotic analgesics within 24 hours prior to enrollment.
   2. Diaminodiphenyl sulfone within 1 week prior to enrollment or etanercept within 2 weeks prior to enrollment.
   3. Intraarticular, intramuscular, or intravenous administration of glucocorticoids within 72h(3 days) prior to enrollment, or intravenous immunoglobulin within 4 weeks prior to enrollment.
   4. Intravenous immunoglobulins with proven Still's disease modifying effect, leflunomide, infliximab, or adalimumab within 8 weeks prior to enrollment.
   5. Thalidomide within 72h(3 days) prior to enrollment, cyclosporine within 5 weeks prior to enrollment, mycophenolate mofetil within 1 week prior to enrollment, 6-mercaptopurine within 48h(2 days) prior to enrollment, azathioprine within 72h(3 days) prior to enrollment, cyclophosphamide within 96h(4 days) prior to enrollment, chlorambucil (not approved inJapan) within 48h(2 days) prior to enrollment, or any other immunosuppressants within 12 weeks prior to enrollment.
   6. Tocilizumab within 4 weeks prior to enrollment or any other immunomodulatory medications within 4 half-lives prior to enrollment.
   7. Rituximab within 13 weeks prior to enrollment.
   8. Canakinumab within 130 days prior to enrollment
3. Live vaccines within 4 weeks prior to enrollment.
4. Known presence or suspicion of active, chronic, or recurrent bacterial, fungal, or viral infections, including but not limited to tuberculosis, HIV infection, Covid-19 infection, or hepatitis B or C infection at baseline. Patients with acute or chronic HBV.
5. Clinical evidence of liver disease or liver injury as indicated by presence of abnormal liver tests.
6. Presence of severe chronic kidney disease (CKD) grades 4 and 5.
7. Presence of neutropenia (absolute neutrophil count [ANC] < 1.5 x 10^9/L).
8. Presence of thrombocytopenia (platelets count < 100 x 10^9/L).
9. Presence or suspicion of MAS at baseline.
10. History or diagnosis of MAS within the last 4 weeks prior to enrollment.

After completion of the study Core Phase, patients who consent and are eligible to continue anakinra treatment, can enter the extension phase .

Min Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
An improvement of ≥ 30% from baseline in physician global assessment of disease activity (visual analogue scale [VAS]). | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days
An improvement of ≥ 30% from baseline in patient/parent global assessment of overall well-being (VAS). | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days
An improvement of ≥ 30% from baseline in number of joints with active arthritis. | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days
An improvement of ≥ 30% from baseline in number of joints with limitation of motion. | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days
An improvement of ≥ 30% from baseline in assessment of physical function: Child health assessment questionnaire (CHAQ)/Stanford health assessment questionnaire (SHAQ). | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days
An improvement of ≥ 30% from baseline in C-reactive protein (CRP) (mg/L). | Week 2
  ACR30 response with absence of fever attributable to the disease during the 7 days

SECONDARY OUTCOMES:
Change in CRP. | Week 2
  To demonstrate the efficacy of anakinra compared to placebo in reducing inflammation in Still's disease.
Change in ferritin. | Week 2
  To demonstrate the efficacy of anakinra compared to placebo in reducing inflammation in Still's disease.
Change in haemoglobin. | Week 2
  To demonstrate the efficacy of anakinra compared to placebo in reducing inflammation in Still's disease.
Change in platelets count. | Week 2
  To demonstrate the efficacy of anakinra compared to placebo in reducing inflammation in Still's disease.
Change in white blood cells count. | Week 2
  To demonstrate the efficacy of anakinra compared to placebo in reducing inflammation in Still's disease.
Absence of fever during the 24 hours preceding the evaluation visit at Week 1. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Absence of rash during the 24 hours preceding the evaluation visit at Week 1. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
ACR30 response with absence of fever during the 24 hours preceding the evaluation visit at Week 1. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
ACR50 response with absence of fever during the 24 hours preceding the evaluation visit at Week 1. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
ACR70 response with absence of fever during the 24 hours preceding the evaluation visit at Week 1. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in physician global assessment of disease activity, measured on a VAS from no pain (0 mm) to very severe (100 mm). | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in patient/parent global assessment of overall well-being, measured on a VAS from no pain (0 mm) to very severe (100 mm). | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in patient/parent global assessment of disease related pain, measured on a VAS from no pain (0 mm) to very severe (100 mm). | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in swelling joints count. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in tender joints count. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in CRP. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in ferritin. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in haemoglobin. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in platelets count. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in white blood cells count. | Week 1
  To demonstrate early onset of efficacy of anakinra compared to placebo in Still's disease.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-Y Proxy (4-7 years). | Week 2
  To evaluate and compare the health status between anakinra treated patients and patients treated with placebo.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-Y (8-15 years). | Week 2
  To evaluate and compare the health status between anakinra treated patients and patients treated with placebo.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-3L (≥ 16 years). | Week 2
  To evaluate and compare the health status between anakinra treated patients and patients treated with placebo.
Absence of fever during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Absence of rash during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
ACR30 response with absence of fever during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
ACR50 response with absence of fever during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
ACR70 response with absence of fever during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
ACR90 response with absence of fever during the 7 days preceding the visit. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in physician global assessment of disease activity (VAS). | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in patient/parent global assessment of overall well-being (VAS). | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in patient/parent global assessment of disease related pain (VAS). | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in swelling joints count. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in tender joints count. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in CRP. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in ferritin. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in haemoglobin. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in platelets count. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Change in white blood cells count. | Week 4 to Week 54
  To evaluate efficacy of anakinra in Still's disease.
Occurrence of inactive disease. | Week 8 to Week 54
  Proportion of patients who reach inactive disease.Inactive disease is defined as no joints with active arthritis, no fever, no rash, serositis, no hepatosplenomegaly, no generalized lymphadenopathy attributable to Still's disease, CRP level within normal limits, physician's global assessment of disease activity score below 10 mm on a 100 mm VAS, and a documented morning stiffness ≤15 min.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-Y Proxy (4-7 years). | Week 4 to Week 54
  To evaluate the health status in anakinra treated patients with Still's disease.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-Y (8-15 years). | Week 4 to Week 54
  To evaluate the health status in anakinra treated patients with Still's disease.
Change in the number/proportion of patients reporting problems by dimension of EQ-5D-3L(≥ 16 years). | Week 4 to Week 54
  To evaluate the health status in anakinra treated patients with Still's disease.
ACR30 response with absence of fever during the 7 days preceding the study visits over time. | Week 2 to Week 54
  To evaluate sustained efficacy of anakinra in patients responding to study drug.
To evaluate the occurrence of study drug discontinuation in anakinra treated patients with Still's disease. | Day 1 to Week 54
  * Time to study drug discontinuation due to lack of efficacy or progressive disease.
  * Time to study drug discontinuation due to any reason.
  * Number of patients discontinuing study treatment.
Time of initiation of glucocorticoids tapering. | Week 2 to Week 54
  To evaluate glucocorticoids tapering in anakinra treated patients with Still's disease.
Percentage decrease of glucocorticoids dose for patients tapering their glucocorticoids dose. | Week 2 to Week 54
  To evaluate glucocorticoids tapering in anakinra treated patients with Still's disease.
Discontinuation of glucocorticoids. | Week 2 to Week 54
  To evaluate glucocorticoids tapering in anakinra treated patients with Still's disease.
- Occurrence of adverse events (AEs) (serious adverse events [SAEs] and non-SAEs). | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
Occurrence of deaths | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
Occurrence of AEs leading to study drug discontinuation at all study visits. | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
Occurrence of vital signs changes from baseline, including blood pressure, heart rate, and body weight at all study visits up to Week 58 visit. Changes of height in patients younger than 19 years old. | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
Occurrence of laboratory safety assessments changes over time. | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
Occurrence of abnormal laboratory values. | Baseline to Week 58
  To evaluate the safety of anakinra in patients with Still ́s disease.
To evaluate immunogenicity of anakinra in patients with Still's disease. | Baseline, Weeks 2, 4, 12, 34, 54 and 58
  * Occurrence of ADAs, NAbs, cross-reactivity, and titer levels of ADAs and NAbs
  * Occurrence and titer levels of ADAs in relation to AEs
  * Occurrence and titer levels of ADAs, NAbs cross-reactivityin relation to ACR30 response and CRP levels
To evaluate the pharmacokinetic of anakinra in patients with Still's disease | Baseline, Weeks 1 and 2
  Anakinra serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Mori, MD, Principal Investigator — St. Marianna University Hospital
Locations (8):
- Japan (8):
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Hospital (Hematology and Clinical Immunology), Yokohama, Kanagawa
  - Shinshu University, Matsumoto, Nagano
  - Tokyo Medical And Dental University Hospital, Bunkyō-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Gifu University Hospital, Gifu

IPD SHARING:
Plan to Share IPD: No